CLINICAL TRIAL: NCT03137108
Title: Effects of Transcutaneous Spinal Cord Stimulation on Residual Voluntary Motor Control, Standing, and Overground Walking in Individuals With Incomplete Spinal Cord Injury Single Centre Pilot Study Investigating Immediate Effects of Transcutaneous Electrical Spinal Cord Stimulation on Voluntary Ankle and Knee Control, Standing and Overground Walking in Incomplete Spinal Cord Injury
Brief Title: Effects of Transcutaneous Spinal Cord Stimulation on Residual Voluntary Motor Control in Individuals With Incomplete Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-00053
Record Dates: First submitted 2017-04-21; First posted 2017-05-02 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Motor Control in Incomplete Spinal Cord Injured Persons

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Incomplete Spinal cord injury (Experimental)
  Interventions: Device: Transcutaneous electrical spinal cord stimulation

INTERVENTIONS:
Device: Transcutaneous electrical spinal cord stimulation — Study intervention consists of the application of tSCS at three different frequencies (15 Hz, 30 Hz, 50 Hz) using the CE certified electrostimulator RehaMove 3. Stimulation will only be applied by an investigator during the two testing sessions. During the overground walking, the participants will be secured and assisted with the cable-driven body-weight support system FLOAT.

SUMMARY:
Recently, a transcutaneous protocol of electrical spinal cord stimulation (tSCS) has been developed. It was suggested, that this method could be used to improve the therapy process after a spinal cord injury (SCI). The aim of this study is to investigate the immediate effects of tSCS with different stimulation modalities on voluntary motor control in patients with incomplete SCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with incomplete SCI
* Chronic (≥ 12 months post-injury) or subacute (≥ 3 months post-injury) stage of recovery
* Age: ≥18 years
* Able to complete the 10mWT with walking aids as required but no physical assistance
* Neurological level of SCI: above T12
* Preserved segmental and cutaneo-muscular reflexes in the lower limbs
* Bodyweight > 20 kg and < 120 kg
* Mini-Mental state examination score 6 (test only performed if cognitive deficits are suspected)

Exclusion Criteria:

* Any other neurological diseases
* Current orthopedic problems
* Premorbid major depression or psychosis
* History of significant autonomic dysreflexia with treatment
* Dermatological issues (e.g. decubitus) at the stimulation or harness attachment site (back, abdomen, upper legs)
* Active implants (e.g. cardiac pacemaker, implanted drug pump)
* Passive implants at vertebral level T9 or more caudal vertebrae (metal screws and plates for surgical stabilization of spinal fractures)
* Malignant diseases
* Heart insufficiency NYHA III-IV
* Potential pregnancy (pregnancy test must be conducted before each session)
* Unlikely to complete the intervention or return for follow-up
* Participation in another training study
* Contraindications for BWS training using the FLOAT (according the manual):
* No responsiveness
* Severe muscle contractures
* Acute fractures
* Osteoporosis or osteogenesis imperfecta
* Body size shorter than 1 meter or taller than 2 meters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Kinematic movement characteristics recorded with a motion capture system; | Baseline and intervention of a specific task will be assessed directly after each other in a single session. All movement tasks will be split into 2 sessions within 2 weeks. The start of the first session is variable.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinik Balgrist, Zurich, Switzerland